CLINICAL TRIAL: NCT01408173
Title: A Phase III Clinical Study of NPC-11 in the Treatment of Apnea of Prematurity. - Investigation of Safety, Efficacy and Pharmacokinetics of Caffeine Citrate -
Brief Title: Clinical Study of Caffeine for Apnea of Prematurity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nobelpharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPC-11-1
Record Dates: First submitted 2011-07-29; First posted 2011-08-03 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-10

CONDITIONS: Apnea of Prematurity
Keywords: caffeine; apnea; prematurity
MeSH Terms: conditions — Apnea; Premature Birth | interventions — Administration, Oral; caffeine citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NPC-11 (Experimental): * Loading Dose (Day 1): Caffeine citrate 20 mg/kg body weight will be administered intravenously using a syringe infusion pump over 30 minutes.
  * Maintenance Dose (Day 2～Day 10): After an interval 24 hours, caffeine citrate 5 mg/kg body weight will be administered intravenously (over 10 minutes) or orally if the patients will be able to receive oral administration once a day. The maintenance dose can be increased to a maximum 10 mg/kg caffeine citrate once a day if apnea persists.
  Interventions: Drug: NPC-11 for intravenous or oral administration.

INTERVENTIONS:
Drug: NPC-11 for intravenous or oral administration. — NPC-11, Each vial (3mL) contains 60 mg caffeine citrate (equivalent to 30mg caffeine).
  Other Names: caffeine citrate

SUMMARY:
The aim of the present Phase III study is to evaluate the safety, efficacy and pharmacokinetics of Caffeine Citrate for treatment of apnea of prematurity in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Postconceptional age between 28 weeks and 33 weeks, and over 24 hours after birth.
* At least 6 episodes of apnea (>20 seconds in duration) in 24 hours.
* Signed written informed consent from parent(s) or legal guardian(s).

Exclusion Criteria:

* Apnea due to: hypoxic-ischemic encephalopathy, meningitis, seizures, Grade III or IV intracranial hemorrhage, CNS depression from drugs administered to the mother during delivery, periventricular leukomalacia, pneumonia which does not improve even if it treats, hemoglobin< 10 g/dL, sepsis, shock which does not improve even if it treats, blood pH<7.2 on 2 consecutive determinations in spite of correction, serum calcium concentration <7.0 mg/dL which does not improve even if it treats, serum glucose concentration <4.0 mg/dL which does not improve even if it treats, congestive heart failure, symptomatic patent ductus arteriosus, rectal temperature>38.5 °C on 2 consecutive readings, rectal temperature< 35 °C on 2 consecutive readings, obstructive apnea.
* Blood urea nitrogen >20 mg/dL, serum creatinine >1.5 mg/dL.
* Serum AST or ALT >3 times the upper limit of normal.
* Requirement of mechanically-assisted ventilation ( containing nasal CPAP, nasal DPAP).
* Previous treatment with methylxanthines within 7 days prior to study enrollment.
* Previous treatment with H2 antagonists (i.e., cimetidine or ranitidine) within 7 days prior to study enrollment.
* Receiving or experiencing the effects of CNS-active medication at the time of enrollment.
* Participant of other clinical trial within 6 months.
* Inappropriate to enter this clinical trial judged by the investigator in charge.

Ages: 28 Weeks to 33 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2011-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Success rates for controlling of apnea episode in each observation day (at least 50% reduction of apnea episodes from baseline) | 1, 2, 3, 4, 5, 6,7, 8, 9 and 10 day

SECONDARY OUTCOMES:
The change of frequency of apnea episode from baseline in each observation day | 1, 2, 3, 4, 5, 6, 7, 8, 9 and 10 day
Time to event：Days until next events occurred | 1 to 10 day
  Time to event：Days until next events occurred.
  The definition of events are, Not at least 50% reduction of apnea episode Not improving the frequency of episode from baseline Needs mechanical/bag valve mask ventilation.
The change of average duration time of apnea episode from baseline in each observation day | 1, 2, 3, 4, 5, 6, 7, 8, 9 and 10 day
The change of lowest oxygen saturation during apnea episodes from baseline in each observation day | 1, 2, 3, 4, 5, 6, 7, 8, 9 and 10 day
The proportion of less than 85% oxygen saturation during apnea episodes in each observation day | 1, 2, 3, 4, 5, 6, 7, 8, 9 and 10 day

CONTACTS AND LOCATIONS:
Overall Officials: Susumu Itoh, MD, PhD, Principal Investigator — Kagawa University
Locations (3):
- Japan (3):
  - Fujita Health University Hospital, Kutsukake, Aichi-ken
  - Osaka Medical Center and Research Institute for Maternal and Child Health, Izumi, Osaka
  - Tokyo Metropolitan Children's Medical Center, Fuchū, Tokyo